CLINICAL TRIAL: NCT02226003
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of the Initial Combination of Ertugliflozin (MK-8835/PF-04971729) With Sitagliptin in the Treatment of Subjects With T2DM With Inadequate Glycemic Control on Diet and Exercise
Brief Title: Efficacy and Safety of Ertugliflozin (MK-8835/PF-04971729) With Sitagliptin in the Treatment of Participants With Type 2 Diabetes Mellitus (T2DM) With Inadequate Glycemic Control on Diet and Exercise (MK-8835-017)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-017; 2014-001049-25 (EudraCT Number); B1521047 (Other: Pfizer Protocol Number)
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin; Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ertugliflozin 5 mg and Sitagliptin 100 mg (Experimental): Ertugliflozin, 5 mg, administered orally, once daily for 26 weeks. Sitagliptin, 100 mg, administered orally, once daily for 26 weeks. Placebo to ertugliflozin, 10 mg, administered orally, once daily for 26 weeks.
  Interventions: Drug: Ertugliflozin; Drug: Sitagliptin; Drug: Placebo to Ertugliflozin; Drug: Glimepiride
- Ertugliflozin 15 mg and Sitagliptin 100 mg (Experimental): Ertugliflozin, 15 mg, administered orally, once daily for 26 weeks. Sitagliptin, 100 mg, administered orally, once daily for 26 weeks.
  Interventions: Drug: Ertugliflozin; Drug: Sitagliptin; Drug: Glimepiride
- Placebo to Ertugliflozin and Placebo to Sitagliptin (Placebo Comparator): Placebo to ertugliflozin, 5 mg and 10 mg, administered orally, once daily for 26 weeks. Placebo to sitagliptin, 100 mg, administered orally, once daily for 26 weeks.
  Interventions: Drug: Placebo to Ertugliflozin; Drug: Placebo to Sitagliptin; Drug: Glimepiride

INTERVENTIONS:
Drug: Ertugliflozin — Ertugliflozin, 5 mg or 15 mg, administered orally, once daily for 26 weeks.
  Arms: Ertugliflozin 15 mg and Sitagliptin 100 mg; Ertugliflozin 5 mg and Sitagliptin 100 mg
Drug: Sitagliptin — Sitagliptin, 100 mg, administered orally, once daily for 26 weeks.
  Arms: Ertugliflozin 15 mg and Sitagliptin 100 mg; Ertugliflozin 5 mg and Sitagliptin 100 mg
Drug: Placebo to Ertugliflozin — Matching placebo to ertugliflozin administered orally, once daily for 26 weeks.
  Arms: Ertugliflozin 5 mg and Sitagliptin 100 mg; Placebo to Ertugliflozin and Placebo to Sitagliptin
Drug: Placebo to Sitagliptin — Matching placebo to sitagliptin administered orally, once daily for 26 weeks.
  Arms: Placebo to Ertugliflozin and Placebo to Sitagliptin
Drug: Glimepiride — Open-label glimepiride rescue therapy will be initiated at 1 or 2 mg/day and may be titrated to the maximum labeled dose or maximum tolerated dose (if lower than labeled dose), as considered appropriate by the investigator, based on blood glucose measurements and in accordance with the local, approved label.

SUMMARY:
This is a study to evaluate the efficacy and safety of ertugliflozin (MK-8835/PF-04971729) in combination with sitagliptin in the treatment of participants with Type 2 diabetes mellitus (T2DM) with inadequate glycemic control on diet and exercise. The primary hypothesis of the study is that ertugliflozin plus sitagliptin is more effective in lowering of hemoglobin A1C (HbA1C) than placebo.

DETAILED DESCRIPTION:
Each participant will be in the study for approximately 39 weeks including: a 1-week screening period, an 8-week (or greater) antihyperglycemic agent (AHA) wash-off period, a 2-week single-blind placebo run-in period, a 26-week double-blind treatment period, and a post-treatment telephone contact 14 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus as per American Diabetes Association guidelines
* Not on antihyperglycemic agent (AHA) >=8 weeks with a Visit 1/Screening HbA1C >=8.0% and <=10.5% (>=64 mmol/mol and <=91 mmol/mol) OR on single allowable AHA (allowable AHAs prior to screening are: metformin, α-glucosidase inhibitors, sulfonylureas and glinides) with a Visit 1/Screening HbA1C >=7.5% and <=10.0% (>=58 mmol/mol and <=86 mmol/mol) OR on low-dose dual combination therapy (≤50% of maximum labeled dose of an AHA) with allowable AHAs with a Visit 1/Screening HbA1C >=7.5% and <=10.0% (>=58 mmol/mol and <=86 mmol/mol)
* Body mass index (BMI) >=18.0 kg/m^2
* Male or female not of reproductive potential
* Female of reproductive potential who agrees to (or have their partner agree to) remain abstinent from heterosexual activity or to use 2 acceptable combinations of contraception.

Exclusion Criteria:

* History of type 1 diabetes mellitus or diabetic ketoacidosis
* History of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant
* A known hypersensitivity or intolerance to any sodium glucose co-transporter (SGLT2) inhibitor or sitagliptin
* Has been treated with any of the following agents within 12 weeks of study start or during the pre-randomization period: insulin of any type (except for short-term use [i.e., <=7 days] during concomitant illness or other stress), other injectable anti-hyperglycemic agents (e.g., pramlintide, exenatide, liraglutide), pioglitazone or rosiglitazone, other sodium glucose co-transporter 2 (SGLT2) inhibitors, dipeptidyl-peptidase 4 inhibitors (DPP-4 inhibitors), bromocriptine (Cycloset™), colesevelam (Welchol™), any other AHA with the exception of the protocol-approved agents
* Is on a weight-loss program or weight-loss medication or other medication associated with weight changes and is not weight stable prior to study start
* Has undergone bariatric surgery within the past 12 months or >12 months and is not weight stable prior to study start
* A history of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, or New York Heart Association (NYHA) functional Class III-IV heart failure within 3 months of study start
* Active, obstructive uropathy or indwelling urinary catheter
* History of malignancy <=5 years prior to study start, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* A known history of human immunodeficiency virus (HIV)
* A blood dyscrasia or any disorder causing hemolysis or unstable red blood cells, or a clinically important hematological disorder (e.g. aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* A medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Any clinically significant malabsorption condition
* Current treatment for hyperthyroidism
* On thyroid replacement therapy and not on a stable dose for at least 6 weeks prior study start
* On a previous clinical study with ertugliflozin
* Participated in other studies involving investigational drug(s) 30 days prior to study start
* Surgical procedure within 6 weeks prior to study start or major surgery planned during the trial
* Positive urine pregnancy test
* Pregnant or breast-feeding, or planning to conceive during the trial, including 14 days following the last dose of study medication
* Planning to undergo hormonal therapy in preparation for egg donation during the trial, including 14 days following the last dose of study medication
* Routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week or engages in binge drinking
* Donated blood or blood products within 6 weeks of study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2016-02-23 (Actual); Study Completion 2016-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Miller S, Krumins T, Zhou H, Huyck S, Johnson J, Golm G, Terra SG, Mancuso JP, Engel SS, Lauring B. Ertugliflozin and Sitagliptin Co-initiation in Patients with Type 2 Diabetes: The VERTIS SITA Randomized Study. Diabetes Ther. 2018 Feb;9(1):253-268. doi: 10.1007/s13300-017-0358-0. Epub 2018 Jan 8. PMID 29313282
- [Derived] Gallo S, Raji A, Calle RA, Pong A, Meyer C. The effects of ertugliflozin on beta-cell function: Pooled analysis from four phase 3 randomized controlled studies. Diabetes Obes Metab. 2020 Dec;22(12):2267-2275. doi: 10.1111/dom.14149. Epub 2020 Aug 27. PMID 32700393
- [Derived] Gallo S, Calle RA, Terra SG, Pong A, Tarasenko L, Raji A. Effects of Ertugliflozin on Liver Enzymes in Patients with Type 2 Diabetes: A Post-Hoc Pooled Analysis of Phase 3 Trials. Diabetes Ther. 2020 Aug;11(8):1849-1860. doi: 10.1007/s13300-020-00867-1. Epub 2020 Jul 9. PMID 32648108
- [Derived] Patel S, Hickman A, Frederich R, Johnson S, Huyck S, Mancuso JP, Gantz I, Terra SG. Safety of Ertugliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Seven Phase 3 Randomized Controlled Trials. Diabetes Ther. 2020 Jun;11(6):1347-1367. doi: 10.1007/s13300-020-00803-3. Epub 2020 May 5. PMID 32372382
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Wu L, Patel S, Hickman A, Mancuso JP, Gantz I, Terra SG. Efficacy and safety of ertugliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Aug;36(8):1277-1284. doi: 10.1080/03007995.2020.1760228. Epub 2020 May 13. PMID 32324082
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Patel S, Hickman A, Mancuso JP, Ellison MC, Gantz I, Terra SG. Efficacy and safety of ertugliflozin in Hispanic/Latino patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Jul;36(7):1097-1106. doi: 10.1080/03007995.2020.1760227. Epub 2020 May 13. PMID 32324065
- [Derived] Liu J, Patel S, Cater NB, Wu L, Huyck S, Terra SG, Hickman A, Darekar A, Pong A, Gantz I. Efficacy and safety of ertugliflozin in East/Southeast Asian patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2020 Apr;22(4):574-582. doi: 10.1111/dom.13931. Epub 2020 Jan 3. PMID 31797522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 96 sites received independent ethics committees/institutional review boards' approval and 66 sites in 9 countries enrolled at least 1 participant.
Pre-assignment Details: The study included a 1-week screening period; an 8-week (or greater) antihyperglycemic agent (AHA) wash-off period; and a 2-week single-blind placebo run-in period.
Groups:
- Ertugliflozin 5 mg + Sitagliptin 100 mg: Ertugliflozin, 5 mg, administered orally, once daily for 26 weeks. Sitagliptin, 100 mg, administered orally, once daily for 26 weeks. Placebo to ertugliflozin, 10 mg, administered orally, once daily for 26 weeks.
- Ertugliflozin 15 mg + Sitagliptin 100 mg: Ertugliflozin, 15 mg, administered orally, once daily for 26 weeks. Sitagliptin, 100 mg, administered orally, once daily for 26 weeks.
- Placebo: Placebo to ertugliflozin, 5 mg and 10 mg, administered orally, once daily for 26 weeks. Placebo to sitagliptin, 100 mg, administered orally, once daily for 26 weeks.
Period: Overall Study
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Started | 98 | 96 | 97
Completed | 96 | 95 | 91
Not Completed | 2 | 1 | 6
Not completed — Lost to Follow-up | 2 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo | Total
Number analyzed (Participants) | 98 | 96 | 97 | 291
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.4 (9.3) | 56.1 (10.1) | 54.3 (10.3) | 55.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 40 | 124
  Male | 57 | 53 | 57 | 167

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (HbA1C) at Week 26 - Full Analysis Set (FAS Population Excluding Rescue Approach
Description: HbA1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). HbA1C represents the percentage of glycated hemoglobin. A negative number indicates a reduction in HbA1C level. Excluding rescue approach excludes all data following the initiation of rescue, in order to avoid the confounding influence of the rescue therapy with open-label glimepiride.
Time Frame: Baseline and Week 26
Population: FAS population includes randomized participants who took at least 1 dose of study medication and had at least one assessment at or after baseline for the change from baseline in the Week 26 HbA1C endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 98 | 96 | 96
Percentage | -1.60 [-1.82 to -1.39] | -1.68 [-1.90 to -1.46] | -0.44 [-0.69 to -0.19]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -1.16, 95% CI 2-sided [-1.49 to -0.84]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -1.24, 95% CI 2-sided [-1.57 to -0.91]

2. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE) - All Participants as Treated Excluding Rescue Approach
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Excluding rescue approach excludes all data following the initiation of rescue, in order to avoid the confounding influence of the rescue therapy with open-label glimepiride.
Time Frame: Up to Week 28
Population: All Subjects as Treated (ASaT) population consisted of all randomized participants who received at least one dose of a study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 98 | 96 | 97
Percentage of Participants | 44.9 | 44.8 | 42.3
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; Difference in Percentage vs Placebo = 2.6, 95% CI 2-sided [-11.2 to 16.4]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; Difference in Percentage vs Placebo = 2.5, 95% CI 2-sided [-11.4 to 16.4]

3. Primary Outcome: Percentage of Participants Who Discontinued Study Medication Due to an AE - All Participants as Treated Excluding Rescue Approach
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Excluding rescue approach excludes all data following the initiation of rescue, in order to avoid the confounding influence of the rescue therapy with open-label glimepiride.
Time Frame: Up to Week 26
Population: ASaT population consisted of all randomized participants who received at least one dose of a study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 98 | 96 | 97
Percentage of Participants | 2.0 | 2.1 | 2.1

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26 - Full Analysis Set Excluding Rescue Approach
Description: Blood glucose was measured after a ≥10 hour fast. Blood was drawn at predose on Day 1 and after 26 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 26 minus FPG at baseline). Excluding rescue approach excludes all data following the initiation of rescue, in order to avoid the confounding influence of the rescue therapy with open-label glimepiride.
Time Frame: Baseline and Week 26
Population: FAS population includes randomized participants who took at least 1 dose of study medication and had at least one assessment at or after baseline for the change from baseline in the Week 26 FPG endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams/deciliter
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 98 | 96 | 96
milligrams/deciliter | -48.25 [-56.12 to -40.38] | -55.36 [-63.29 to -47.42] | -9.30 [-18.58 to -0.02]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -38.94, 95% CI 2-sided [-49.93 to -27.96]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -46.05, 95% CI 2-sided [-57.09 to -35.02]

5. Secondary Outcome: Change From Baseline in 2-hour Post-Meal Glucose (PMG) at Week 26 - Full Analysis Set Excluding Rescue Approach
Description: Change from baseline at Week 26 is defined as 2-hour PMG at Week 26 minus 2-hour PMG at Week 0. Two-hour post-meal glucose was measured following a standard meal. Excluding rescue approach excludes all data following the initiation of rescue, in order to avoid the confounding influence of the rescue therapy with open-label glimepiride.
Time Frame: Baseline and Week 26
Population: FAS population is all randomized participants who took at least 1 dose of study medication and had at least one assessment at or after baseline for the change from baseline in the Week 26 2-hour PMG endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams/deciliter
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 97 | 95 | 91
milligrams/deciliter | -82.80 [-95.96 to -69.64] | -90.03 [-103.34 to -76.71] | -20.38 [-35.62 to -5.14]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -62.42, 95% CI 2-sided [-80.47 to -44.37]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -69.65, 95% CI 2-sided [-87.83 to -51.46]

6. Secondary Outcome: Percentage of Participants With HbA1C <7% (<53 mmol/Mol) at Week 26
Description: HbA1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). HbA1c represents the percentage of glycated hemoglobin.
Time Frame: Week 26
Population: FAS population includes randomized participants who took at least 1 dose of study medication and had at least one assessment at or after baseline in the Week 26 HbA1C endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 98 | 96 | 96
Percentage of participants | 35.7 | 31.3 | 8.3
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Logistic regression model; Odds Ratio (OR) = 6.88, 95% CI 2-sided [2.81 to 16.83]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Logistic regression model; Odds Ratio (OR) = 7.39, 95% CI 2-sided [2.98 to 18.31]

7. Secondary Outcome: Change From Baseline in Body Weight at Week 26 - Full Analysis Set Excluding Rescue Approach
Description: Body weight was measured using a standardized, digital scale at each of the pre-defined nominal time points. Weight was taken in duplicate throughout the trial at approximately the same time of day, after voiding (i.e., forced void) and while wearing only a gown and underwear. Excluding rescue approach excludes all data following the initiation of rescue, in order to avoid the confounding influence of the rescue therapy with open-label glimepiride.
Time Frame: Baseline and Week 26
Population: FAS population is all randomized participants who took at least 1 dose of study medication and had at least one assessment at or after baseline for the change from baseline in the Week 26 body weight endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 98 | 96 | 97
Kilograms | -2.94 [-3.60 to -2.28] | -3.04 [-3.71 to -2.38] | -0.94 [-1.70 to -0.18]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -2.00, 95% CI 2-sided [-2.99 to -1.01]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -2.10, 95% CI 2-sided [-3.10 to -1.11]

8. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure at Week 26 - Full Analysis Set Excluding Rescue Approach
Description: Blood pressure measurements were taken after at least 5 minutes of rest. Three measurements were taken approximately 2 minutes apart with the triplicate set recorded. Excluding rescue approach excludes all data following the initiation of rescue, in order to avoid the confounding influence of the rescue therapy with open-label glimepiride.
Time Frame: Baseline and Week 26
Population: FAS population included all randomized participants who took at least 1 dose of study medication and had at least one assessment at or after baseline for the change from baseline in the Week 26 sitting systolic blood pressure endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters of mercury
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 98 | 96 | 97
millimeters of mercury | -2.04 [-4.23 to 0.16] | -3.98 [-6.19 to -1.78] | 2.41 [-0.34 to 5.15]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p = 0.011, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -4.44, 95% CI 2-sided [-7.87 to -1.01]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -6.39, 95% CI 2-sided [-9.83 to -2.95]

9. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure at Week 26 - Full Analysis Set Excluding Rescue Approach
Description: as for outcome 8
Time Frame: Baseline and Week 26
Population: The FAS population included all randomized participants who took at least 1 dose of study medication and had at least one assessment at or after baseline for the change from baseline in the Week 26 sitting diastolic blood pressure endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters of mercury
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 98 | 96 | 97
millimeters of mercury | -0.44 [-1.99 to 1.11] | -0.97 [-2.52 to 0.59] | 1.21 [-0.73 to 3.15]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p = 0.184, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -1.65, 95% CI 2-sided [-4.09 to 0.79]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg + Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p = 0.080, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -2.18, 95% CI 2-sided [-4.62 to 0.26]

ADVERSE EVENTS:
Time Frame: Up to Week 28
Description: The serious adverse event table includes events after the initiation of glycemic rescue. The non-serious adverse event table excludes events after the initiation of glycemic rescue.
Arm/Group | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/98 | 3/96 | 5/97
Other Adverse Events (participants affected / at risk) | 8/98 | 3/96 | 12/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg + Sitagliptin 100 mg (N=98) | Ertugliflozin 15 mg + Sitagliptin 100 mg (N=96) | Placebo (N=97)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg + Sitagliptin 100 mg (N=98) | Ertugliflozin 15 mg + Sitagliptin 100 mg (N=96) | Placebo (N=97)
Blood glucose increased (Investigations) | 3 (4) | 0 (0) | 7 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (6)
Urinary tract infection (Infections and infestations) | 5 (6) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.